CLINICAL TRIAL: NCT07359859
Title: Randomized Pilot Study of Ruxolitinib for Switch-Maintenance Prophylaxis of Graft-versus-Host Disease in Allogeneic Hematopoietic Cell Transplantation After Intermediate-Dose Post-Transplant Cyclophosphamide (Rux Switch-Maintenance in Intermediate PTCY: RuSMa-PTCY) in Comparison to Full-Dose PTCY
Brief Title: A Study of Ruxolitinib for Preventing Graft-Versus-Host Disease in People With a Hematologic Malignancy Who Will Receive a Stem Cell Transplant
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-212
Record Dates: First submitted 2026-01-21; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Hematologic Malignancies
Keywords: graft-versus-host disease (GVHD); allogeneic hematopoietic stem cell transplant (allo-HCT)
MeSH Terms: conditions — Hematologic Neoplasms; Graft vs Host Disease | interventions — Cyclophosphamide; Mycophenolic Acid; ruxolitinib; Tacrolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- An intermediate dose (medium dose) of PTCY, tacrolimus, MMF, and the drug ruxolitinib (Experimental): will receive an intermediate (medium) dose of PTCY, tacrolimus, MMF,and ruxolitinib
  Interventions: Drug: Cyclophosphamide; Drug: Mycophenolate Mofetil; Drug: Ruxolitinib; Drug: Tacrolimus
- A full dose of PTCY, tacrolimus, and MMF (the standard GVHD prevention approach) (Active Comparator): will receive a full dose of PTCY, tacrolimus, and MMF (the standard GVHD prevention approach)
  Interventions: Drug: Cyclophosphamide; Drug: Mycophenolate Mofetil; Drug: Tacrolimus

INTERVENTIONS:
Drug: Cyclophosphamide — An intermediate dose (medium dose) of Post-transplant Cyclophosphamide
  Arms: An intermediate dose (medium dose) of PTCY, tacrolimus, MMF, and the drug ruxolitinib
Drug: Cyclophosphamide — A full dose of Post-transplant Cyclophosphamide
  Arms: A full dose of PTCY, tacrolimus, and MMF (the standard GVHD prevention approach)
Drug: Mycophenolate Mofetil — Day +5 to +35
  Other Names: MMF
Drug: Ruxolitinib — twice a day
  Arms: An intermediate dose (medium dose) of PTCY, tacrolimus, MMF, and the drug ruxolitinib
Drug: Tacrolimus — Day +5, taper per SoC
  Arms: A full dose of PTCY, tacrolimus, and MMF (the standard GVHD prevention approach)
Drug: Tacrolimus — Day +5, taper initiation within 2 weeks of starting Ruxolitinib
  Arms: An intermediate dose (medium dose) of PTCY, tacrolimus, MMF, and the drug ruxolitinib

SUMMARY:
The researchers are doing this study to compare 2 different GVHD prevention (prophylaxis) approaches. The researchers will see which approach is good or more effective at preventing chronic GVHD until 1 year after allogeneic hematopoietic stem cell transplantation (allo-HCT).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18- years-old at time of consent
* Diagnosis: hematologic malignancy in morphologic remission (blasts <5%, no evidence of extramedullary disease in AML or MDS). Patients with CR with incomplete count recovery (CRp or CRi) or minimal residual disease are allowed. Patients with lymphoma must have a complete or partial response
* Donor: related or unrelated 7-8/8 HLA-matched or related haploidentical
* Karnofsky score ≥ 70%
* Female subjects of childbearing potential (<50 years old) have a negative serum or urine pregnancy test. Females of childbearing potential are defined as females without prior hysterectomy or who have had any evidence of menses in the past 12 months.

  °Sexually active females of childbearing potential enrolled in the study must agree to consistently use two forms of accepted methods of contraception during the course of the study and for 3 months after their last dose of the study drug. Effective birth control includes: *Intrauterine device (IUD) plus one barrier method *Stable doses of hormonal contraception for at least 3 months (e.g., oral, injectable, implant, transdermal) plus one barrier method *2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gel that contain a chemical to kill sperm); or * A vasectomized partner.
* For male subjects who are sexually active and who are partners of females of childbearing potential: Agreement to use two forms of contraception as per above and to not donate sperm during the treatment period and for at least 3 months after the last dose of study drug

Exclusion Criteria:

* Recipient of CD34+ selected or engineered stem cell graft
* Treatment with in vivo T cell depletion (e.g. anti-thymocyte globulin)
* Severely impaired renal function defined by serum creatinine > 2mg/dL, renal dialysis requirement.
* Use of investigational agent within 14 days pre-HCT
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months
* Uncontrolled psychiatric illness
* Female patient who is pregnant or breastfeeding
* Known allergy or sensitivity to ruxolitinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
assess cGVHD-free survival | 1 year post-HCT
  Chronic GVHD-free survival is defined as moderate-to-severe cGVHD requiring systemic immunosuppression treatment from the date of allo-HCT to first occurrence with follow-up through 12 months post-HCT or death.

SECONDARY OUTCOMES:
incidence of grade 2-4 infections. | 1 year
  Grade 2-4 infections by CTCAE v5 either clinically or microbiologically will be assessed throughout the study until day +365. Causality and relationship with ruxolitinib will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Ponce, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/